CLINICAL TRIAL: NCT01819766
Title: Detection of Advanced Colorectal Neoplasia by Stool DNA in Inflammatory Bowel Disease: OCEANIA Study
Brief Title: Detection of Advanced Colorectal Neoplasia by Stool DNA in Inflammatory Bowel Disease
Acronym: OCEANIA
Status: Completed | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Exact Sciences 2013-01
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2016-08

CONDITIONS: Inflammatory Bowel Disease (IBD); Primary Sclerosing Cholangitis (PSC); Colorectal Neoplasms; Colorectal Cancer
Keywords: Cancer; Colorectal Cancer; Neoplasm; Colorectal Neoplasm; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Inflammatory Bowel Disease; Primary Sclerosing Cholangitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Cholangitis, Sclerosing; Colorectal Neoplasms; Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Residual samples may be archived for further research. Clinical data and samples will be kept in a manner that preserves anonymity of the subject. Specimens will be stored in a commercial biorepository contracted by Exact Sciences or at Exact Sciences and may be used for future research.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IBD or PSC: Subjects will be men and women, 18 to 84 years of age, inclusive, who are at increased risk of developing colorectal cancer.

SUMMARY:
This study aims to determine the performance of the Exact IBD-ACRN surveillance test to detect colorectal cancer (CRC) and colorectal neoplasia in patients with inflammatory bowel disease (IBD). Patients with an IBD diagnosis for at least eight years or diagnosis of primary sclerosing cholangitis (PSC) and who are eligible for CRC screening are eligible to participate in this study. Enrolled subjects will collect a stool sample for the Exact IBD-ACRN surveillance test. Subjects must have undergone colonoscopy no more than 90 days prior to enrollment and will undergo colonoscopy or surgical intervention within 120 days of enrollment. Tissue diagnosis of CRC will be established by histopathologic examination.

DETAILED DESCRIPTION:
This is a prospective, cross sectional, multi-center study to determine the sensitivity and specificity of the Exact IBD-ACRN surveillance test for detecting CRC alone and in combination with high grade dysplasia (HGD) and low grade dysplasia (LGD) associated with IBD and advanced adenoma in IBD patients with disease duration greater than 8 years or PSC diagnosis. Enrolled subjects will provide a single stool sample for the Exact IBD-ACRN surveillance test, no sooner than 7 days following their most recent pre-enrollment colonoscopy, within 30 days of enrollment and prior to initiating bowel prep for either the post-enrollment colonoscopy (surveillance or repeat), or surgical intervention. Stool samples will be tested using the Exact IBD-ACRN surveillance test and results compared to the colonoscopy and corresponding diagnostic histopathology results from biopsied, and any subsequently excised, lesions to establish sensitivity and specificity of the Exact IBD-ACRN surveillance test. All post-enrollment colonoscopies or surgical interventions must be performed within 60 days of enrollment.

The primary objective of this study is to determine the sensitivity and specificity of the Exact IBD-ACRN surveillance test for CRC in IBD patients with disease duration of at least eight years or diagnosis of PSC. Tissue diagnosis of CRC will be established by histopathology examination. The secondary objective is to determine the sensitivity and specificity of the Exact IBD-ACRN surveillance test to detect ACRN in IBD patients with disease duration of at least eight years or diagnosis of PSC.

Enrollment will continue until at least 35 CRC; 15 HGD and 315 negative subject samples have been obtained. There is no specific recruitment goal for IBD associated LGD or LGD associated with advanced adenoma (AA).

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-84 years of age, inclusive.
* Diagnosis of IBD or a diagnosis of PSC with IBD prior to enrollment date of this study.
* Must be a candidate for a surveillance colonoscopy, with the intention of CRC/dysplasia surveillance, or a candidate for surgical intervention based on prior histological confirmation of HGD or CRC.
* Written informed consent document signed and dated by the subject or legally acceptable representative.

Exclusion Criteria:

* Any condition that in the opinion of the investigator should preclude participation in the study.
* A history of aerodigestive tract cancer.
* Prior colorectal resection, except ileocolic resection in Crohn's disease patients.
* IBD limited only to the rectum and without a concurrent PSC diagnosis.
* Subject has participated in any clinical study within the previous 30 days wherein an investigational compound or device was, or may be, introduced into the subject.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have diagnosed IBD and are undergoing a colorectal cancer surveillance program. Also, have either a histopathological diagnosis of high grade dysplasia or colorectal cancer resulting from colonoscopy preceding enrollment or for whom a surveillance colonscopy is indicated.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2013-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the Exact Sciences IBD-ACRN screening test for CRC. | 9 months
  With comparison to the colonoscopy results and histopathologic diagnosis of all lesions discovered during colonoscopy and either biopsied or removed during or subsequently removed after colonoscopy.

SECONDARY OUTCOMES:
Determine Sensitivity and Specificity of the Exact Sciences IBD-ACRN screening test for CRC and HGD. | 9 months
  Subjects with colonoscopic findings of CRC and/or high grade dysplasia (HGD) will be considered to have a positive outcome for composite CRC-HGD sensitivity calculations. Subjects with negative colonoscopic findings will be considered to have a negative outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Itzkowitz, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (26):
- United States (24):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - UC San Diego Medical Center, La Jolla, California
  - University of Miami, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - MGG Group, Co. Inc./Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Detroit Clinical Research Center, PC, Farmington Hills, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Center for Digestive and Liver Diseases, Inc, Mexico, Missouri
  - Mount Sinai School of Medicine, New York, New York
  - Medical Research Associates of New York, New York, New York
  - Asheville Gastroeneterology Associates, Asheville, North Carolina
  - Univeristy of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - Advanced Research Institute, Logan, Utah
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Winnipeg Regional Health Authority-Health Sciences, Winnipeg, Manitoba